CLINICAL TRIAL: NCT04589338
Title: Impact of Different Types of Physical Activity in Patients With Chronic Inflammatory Bowel Disease
Acronym: ACHILLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gofflot Amandine, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20202021
Record Dates: First submitted 2020-09-22; First posted 2020-10-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Diseases; Exercise Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Endurance Training; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endurance training group (Experimental)
  Interventions: Other: Endurance training
- Resistance training group (Experimental)
  Interventions: Other: Resistance training
- Control group (No Intervention)

INTERVENTIONS:
Other: Endurance training — This group will perform aerobic type exercises. Initially, patients will perform continuous exercises of progressive intensity in order to adapt to this kind of effort. Next, we will introduce interval exercises.
  Arms: Endurance training group
Other: Resistance training — Patients in this group will perform lower limb strengthening exercises to improve the maximum strength of different muscle groups.
  Arms: Resistance training group

SUMMARY:
This is a prospective interventional study. The investigators will include patients in clinical remission who are on stable treatment. These IBD patients will be followed to analyze the effects of physical activity on their inflammatory disease. Different exercises will be offered to two separate groups of randomly distributed patients: the first group will perform muscle building exercises while the other group will be offered aerobic exercises.There will also be a control group that does not initially benefit from a specific physical activity program. However, this group will be integrated into one of the other two groups after the 10-week follow-up. All three groups will perform the same baseline tests. These will be of different types: physical tests, biological tests and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients in remission defined by a Harvey Bradshaw Index 5 in Crohn's disease (CD) and a clinical Mayo 3 with no sub-score >1 in ulcerative colitis (RCUH) with stable treatment, without corticosteroid for 4 months.
* Patients accepting the study protocol

Exclusion Criteria:

* Patients suffering from other pathologies (at the level of the digestive system, the cardiovascular system, as well as the musculoskeletal system: recent knee plasty, recent knee fractures, etc.), which can interfere with planned tests and activity programs.
* Patients with more than 3 hours of sports activity per week
* Pregnant, pregnant or nursing patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Progressive effort test on bicycle ergometer (VO2 max) | day 1
  This test allows to measure VO2 in ml/min/kg (thanks to respiratory gases)
Progressive effort test on bicycle ergometer (VO2 max) | through study completion, an average of 40 weeks
  This test allows to measure VO2 in ml/min/kg (thanks to respiratory gases)
Progressive effort test on bicycle ergometer (Heart rate) | day 1
  This test allows to measure resting and maximum heart rate (thanks to an ECG) and maximum aerobic power in Watt.
Progressive effort test on bicycle ergometer (Heart rate) | through study completion, an average of 40 weeks
  This test allows to measure resting and maximum heart rate (thanks to an ECG) and maximum aerobic power in Watt.
Progressive effort test on bicycle ergometer (Power) | day 1
  This test allows to measure maximum aerobic power in Watt.
Progressive effort test on bicycle ergometer (Power) | through study completion, an average of 40 weeks
  This test allows to measure maximum aerobic power in Watt.
Maximum force test (N/m) | Day 1
  This test will be performed using an isokinetic dynamometer. This evaluation will allow us to determine the maximum force of the quadriceps and hamstrings of each participant in N/m.
Maximum force test (N/m) | through study completion, an average of 40 weeks
  This test will be performed using an isokinetic dynamometer. This evaluation will allow us to determine the maximum force of the quadriceps and hamstrings of each participant in N/m.
Blood sample | Day 1
  This type of tests includes biological monitoring to obtain information on biological parameters.
Blood sample | through study completion, an average of 40 weeks
  This type of tests includes biological monitoring to obtain information on biological parameters.
Saddle analysis | Day 1
  This type of tests includes biological monitoring to obtain information on biological parameters.
Saddle analysis | through study completion, an average of 40 weeks
  This type of tests includes biological monitoring to obtain information on biological parameters.
IBD-F | Week 1
  Participants will complete a questionnaire on fatigue perceived.
IBD-F | Week 10
  Participants will complete a questionnaire on fatigue perceived.
IBD-F | Week 20
  Participants will complete a questionnaire on fatigue perceived.
Godin Leisure Time exercise questionnaire | Week 1
  Participants will complete a questionnaire on the level of physical activity
Metabolic Equivalent Task questionnaire | Week 1
  Participants will complete a questionnaire on the level of inactivity
Metabolic Equivalent Task questionnaire | Week 10
  Participants will complete a questionnaire on the level of inactivity
Metabolic Equivalent Task questionnaire | Week 20
  Participants will complete a questionnaire on the level of inactivity
Short Food Frequency Questionnaire | Week 1
  Participants will complete a questionnaire on their dietary habits
Short Food Frequency Questionnaire | Week 10
  Participants will complete a questionnaire on their dietary habits
Short Food Frequency Questionnaire | Week 20
  Participants will complete a questionnaire on their dietary habits
EQ5D questionnaire | Week 1
  Participants will complete a questionnaire on their level of health
EQ5D questionnaire | Week 10
  Participants will complete a questionnaire on their level of health
EQ5D questionnaire | Week 20
  Participants will complete a questionnaire on their level of health
Short health scale questionnaire | Week 1
  Participants will complete a questionnaire to evaluate the level of the inflammatory bowel disease
Short health scale questionnaire | Week 10
  Participants will complete a questionnaire to evaluate the level of the inflammatory bowel disease
Short health scale questionnaire | Week 20
  Participants will complete a questionnaire to evaluate the level of the inflammatory bowel disease

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Liège, Liège, Belgium